CLINICAL TRIAL: NCT00945776
Title: Weekly Phone Calls vs. Brief Patient Education to Improve CPAP Compliance: A Randomized Controlled Trial
Brief Title: Weekly Phone Calls Versus Brief Patient Education to Improve Continuous Positive Airway Pressure (CPAP) Compliance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: George L. Zaldivar, M.D., CAMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-04-2047
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: OSA; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weekly phone calls (Active Comparator): Will be called weekly to answer questions regarding usage.
  Interventions: Behavioral: Weekly phone calls
- Frequently asked questions (Active Comparator): Providing written general answers to commonly asked questions.
  Interventions: Behavioral: Frequently asked questions
- Usual care (Active Comparator)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Weekly phone calls — Calling weekly to answer questions regarding CPAP usage.
  Arms: Weekly phone calls
Behavioral: Frequently asked questions — Answers to frequently asked questions in pre-printed form.
  Arms: Frequently asked questions
Behavioral: Usual care — Answers will be provided by the renter of the equipment, and the sleep center if asked in addition to explanations by the sleep specialist.
  Arms: Usual care

SUMMARY:
The purpose of this study is to compare the effects of three interventions on CPAP adherence.

DETAILED DESCRIPTION:
To determine whether there is a need for a more intensive one on one interaction with the patient in order to improve CPAP usage. And also to try to identify in general which population of patients may require a more intensive intervention.

ELIGIBILITY:
Inclusion Criteria:

* All new patients undergoing of the Sleep Center suspected of having sleep apnea and undergoing sleep studies

Exclusion Criteria:

* Refusal to participate, or not suspected of having sleep apnea prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine which intervention will improve CPAP compliance in sleep apnea | 6 weeks

SECONDARY OUTCOMES:
To try to identify which individual characteristics within a group may require a specific intervention | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George L Zaldivar, M.D., Principal Investigator — CAMC Health System
Locations (1):
- CAMC Sleep Center, Charleston, West Virginia, United States